CLINICAL TRIAL: NCT04644068
Title: A Modular Phase I/IIa, Open-label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of Ascending Doses of AZD5305 as Monotherapy and in Combination With Anti-cancer Agents in Patients With Advanced Solid Malignancies
Brief Title: Study of AZD5305 as Monotherapy and in Combination With Anti-cancer Agents in Patients With Advanced Solid Malignancies
Acronym: PETRA
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D9720C00001; 2020-002688-77 (EudraCT Number)
Record Dates: First submitted 2020-10-26; First posted 2020-11-25 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Ovarian Cancer; Breast Cancer; Pancreatic Cancer; Prostate Cancer; Additional Indications Below for Module 4 and 5; Non-small Cell Lung Cancer; Colorectal Cancer; Bladder Cancer; Gastric Cancer; Biliary Cancer; Cervical Cancer; Endometrial Cancer; Small Cell Lung Cancer Only in Module 5
Keywords: PARP inhibitor; Breast Cancer; Pancreatic Cancer; Prostate Cancer; Ovarian Cancer; AZD5305, T-DXd, Enhertu, Trastuzumab Deruxtecan, Dato-DXd, Datopotamab Deruxtecan, Camizestrant
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Urinary Bladder Neoplasms; Stomach Neoplasms; Biliary Tract Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms | interventions — AZD5305; Paclitaxel; Carboplatin; AZD9833

STUDY DESIGN:
Intervention Model Description: The study consists of individual modules each evaluating the safety and tolerability of AZD5305 dosed as monotherapy, or with a specific combination partner:
  * Module 1 (AZD5305 monotherapy)
  * Module 2 (AZD5305 in combination with paclitaxel)
  * Module 3 (AZD5305 in combination with carboplatin, with or without paclitaxel)
  * Module 4 (AZD5305 in combination with T DXd)
  * Module 5 (AZD5305 in combination with Dato-DXd).
  * Module 6 (AZD5305 in combination with Camizestrant)
  Modules 1 and 4 has 2 study parts: Part A consisting of dose-escalation cohorts and Part B, consisting of expansion cohorts. Modules 2, 3, 5 and 6 have only PART A.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Module 1: AZD5305 Monotherapy (Experimental): AZD5305 Monotherapy
  Interventions: Drug: AZD5305
- Module 2: AZD5305 + Paclitaxel (Experimental): AZD5305 + Paclitaxel
  Interventions: Drug: AZD5305; Drug: Paclitaxel
- Module 3: AZD5305 + Carboplatin with or without Paclitaxel (Experimental): AZD5305 + Carboplatin with or without Paclitaxel
  Interventions: Drug: AZD5305; Drug: Paclitaxel; Drug: Carboplatin
- Module 4: AZD5305 + Trastuzumab Deruxtecan (Experimental): AZD5305 + T- DXd
  Interventions: Drug: AZD5305; Drug: T- Dxd
- Module 5 AZD5305 + Datopotamab Deruxtecan (Experimental): AZD5305 + Dato-DXd
  Interventions: Drug: AZD5305; Drug: Dato-DXd
- Module 6 AZD5305 + Camizestrant (Experimental): AZD5305 + Camizestrant
  Interventions: Drug: AZD5305; Drug: Camizestrant

INTERVENTIONS:
Drug: AZD5305 — Oral PARP inhibitor
Drug: Paclitaxel — IV Anti-microtubule agent
  Arms: Module 2: AZD5305 + Paclitaxel; Module 3: AZD5305 + Carboplatin with or without Paclitaxel
Drug: Carboplatin — IV Platinum chemotherapeutic
  Arms: Module 3: AZD5305 + Carboplatin with or without Paclitaxel
Drug: T- Dxd — IV Antibody-drug conjugate
  Arms: Module 4: AZD5305 + Trastuzumab Deruxtecan
Drug: Dato-DXd — IV Antibody-drug conjugate
  Arms: Module 5 AZD5305 + Datopotamab Deruxtecan
Drug: Camizestrant — Oral SERD Molecule
  Arms: Module 6 AZD5305 + Camizestrant

SUMMARY:
This research is designed to determine if experimental treatment with PARP inhibitor, AZD5305, alone, or in combination with anti-cancer agents is safe, tolerable, and has anti-cancer activity in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study is a Phase I/IIa modular, open-label, multi-center study of AZD5305 administered orally, either as monotherapy or in combination with other anti-cancer agents in patients with advanced solid malignancies.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥ 18 at the time of screening
* Histological or cytological confirmation of advanced malignancy considered to be suitable for study treatment and meeting module specific eligibility criteria..
* Eastern Cooperative Oncology Group Performance status (ECOG PS: 0-2)
* Life expectancy ≥ 12 weeks
* Progressive cancer at the time of study entry
* Patients must have evaluable disease as defined in module-specific criteria for Part A and Part B
* Adequate organ and marrow function as defined by the protocol.
* For Part B expansion cohorts: Provision of formalin-fixed and paraffin embedded (FFPE) tumour specimen is mandatory, where available, except if stated that it is optional in a specific Module.

For Part A:

- Patients may have received up to one prior line of therapy with a PARPi-based regimen (either as a treatment or as maintenance)

For Part B:

- Patients must not have received prior therapy with a PARPi-based regimen (either as a treatment or as maintenance).

Key Exclusion Criteria:

* Treatment with any of the following:

  1. Nitrosourea or mitomycin C within 6 weeks of the first dose of study treatment
  2. Any investigational agents or study drugs from a previous clinical study within 5 half-lives or 3 weeks (whichever is shorter) of the first dose of study treatment
  3. Any other chemotherapy, immunotherapy or anticancer agents within 3 weeks of the first dose of study treatment
  4. Any live virus or bacterial vaccine within 28 days of the first dose of study treatment
* Concomitant use of medications or herbal supplements known to be cytochrome P450 3A4 (CYP3A4) strong inhibitors or inducers.
* Concomitant use of drugs that are known to prolong or shorten QT and have a known risk of Torsades de Pointes.
* Receiving continuous corticosteroids at a dose of >10 mg prednisone/day or equivalent for any reason.
* Major surgery within 4 weeks of the first dose of study treatment.
* Radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of study treatment.
* Any history of persisting (> 2 weeks) severe pancytopenia due to any cause
* Spinal cord compression or brain metastases unless asymptomatic, treated and stable and not requiring continuous corticosteroids at a dose of >10mg prednisone/day or equivalent for at least 4 weeks prior to start of study treatment. Patients with leptomeningeal carcinomatosis are excluded.
* patient with known predisposition to bleeding (e.g., active peptic ulceration, recent [within 6 months] haemorrhagic stroke, proliferative diabetic retinopathy).
* Cardiac conditions as defined by the clinical study protocol
* Other cardiovascular diseases as defined by any of the following:

  1. Symptomatic heart failure,
  2. uncontrolled hypertension,
  3. hypertensive heart disease with significant left ventricular hypertrophy
  4. acute coronary syndrome (ACS)/acute myocardial infarction (AMI), unstable angina pectoris, coronary intervention procedure with percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG) within 6 months.
  5. cardiomyopathy of any etiology
  6. presence of clinically significant valvular heart disease
  7. history of atrial or ventricular arrhythmia requiring treatment; subjects with atrial fibrillation and optimally controlled ventricular rate (< 100 beats per minute) are permitted.
  8. subjects with atrial fibrillation and optimally controlled ventricular rate are permitted
  9. transient ischaemic attack, or stroke within 6 months prior to screening
  10. patients with symptomatic hypotension at screening
* Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of myelodysplastic syndrome (MDS)/acute myeloid leukaemia (AML).
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of AZD5305
* Known allergy or hypersensitivity to investigational product(s) or any of the excipients of the investigational product(s).

Prior malignancy whose natural history, in the Investigator's opinion, has the potential to interfere with safety and efficacy assessments of the investigational regimen.

other module-specific criteria may apply

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 702 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
The number of subjects with adverse events/serious adverse events | From time of Informed Consent to 28 + 7 days post last dose ( modules 1,2,3,5 and 6). 40+7 days post last dose for Module 4.
  Number of patients with adverse events and with serious adverse events including abnormal clinical observations, abnormal ECG parameters, abnormal laboratory assessments and abnormal vital signs that changed from baseline
The number of subjects with dose-limiting toxicity (DLT), as defined in the protocol. | From first dose of study treatment until the end of Cycle 1.
  A DLT is defined as any toxicity that occurs from the first dose of study treatment (either AZD5305 or combination anti-cancer agent) up to and including the planned end of Cycle 1 (the DLT assessment period) that is assessed as unrelated to the disease or disease-related processes under investigation. DLTs occurring outside the DLT window (ie, late onset toxicities) may be defined as a DLT after consultation with the sponsor and investigators, based on the emerging safety profile.

SECONDARY OUTCOMES:
Best percentage change in target lesion | From Screening to confirmed progressive disease (approximately 1 year)
  Change in target lesion size from baseline, as defined by RECIST 1.1.
Objective Response Rate | From Screening to confirmed progressive disease (approximately 1 year)
  Best response until progression, as defined by RECIST 1.1.
Duration of Response | From Screening to confirmed progressive disease (approximately 1 year)
  Time from first response to progression or death , as defined by RECIST 1.1.
Progression Free Survival | From Screening to confirmed progressive disease (approximately 1 year)
  Time from C1D1 to progression or death, as defined by RECIST 1.1.
Time To Response | From Screening to confirmed progressive disease (approximately 1 year)
  Time from C1D1 to complete or partial response, as defined by RECIST 1.1.
Effects of AZD5305 on pH2AX (Ser139) PD biomarker | From Cycle 0 Day 1 to Cycle 1 Day 15 (approximately 21 days)
  Measure change from baseline in pH2AX
CA125 response (ovarian cancer) | From Screening to confirmed progressive disease (approximately 1 year)
  at least a 50% reduction in CA125 levels from a pre-treatment sample as defined by GCIG criteria.
Module 1: Area Under Curve (AUC) | At predefined intervals throughout the treatment period (approximately 12 weeks)
  The concentration of AZD5305 in plasma will be determined. Area under the curve is the integral of the concentration-time curve. The AUC reflects the actual body exposure to drug after administration. The AUC is dependent on the rate of elimination of the drug from the body and the dose administered.
Module 1: Maximum plasma concentration of the drug (Cmax) | At predefined intervals throughout the treatment period (approximately 12 weeks)
  The concentration of AZD5305 in plasma will be determined (Cmax will be derived).
Module 1: The time taken to reach the maximum concentration (Tmax) | At predefined intervals throughout the treatment period (approximately 12 weeks)
  The concentration of AZD5305 in plasma will be determined (Tmax will be derived).
Module 1 and Module 5: Objective Response Rate (prostate cancer) | From Screening to confirmed progressive disease (approximately 1 year)
  Best response until progression, as defined by RECIST 1.1 or PCWG3 (bone)
Module 1: Radiographic progression free survival (prostate cancer) | From Screening to confirmed progressive disease (approximately 1 year)
  Time from C1D1 to progression or death, as defined by RECIST 1.1 and PCWG3(bone).
Module 1: Proportion of subjects with ≥ 50% PSA decrease (prostate cancer) | From Screening to confirmed progressive disease (approximately 1 year)
  PSA from baseline to the lowest post-baseline PSA result, confirmed by a second consecutive PSA assessment
Module 1 : To investigate the effect of a high-fat meal on the PK of AZD5305 | Cycle 0, Day 1 (C0D1), in either the "fasted" or "fed" state, followed by a single oral dose of AZD5305 in the other state for Cycle 1, Day 1 (C1D1) at least 72 hours later; 1 cycle is 28 days.
  Effect on High fat meal on PK parameters of AZD5305.PK parameters, including but not limited to AUC and/or AUC(0-t), Cmax, Tmax, AUC(0-t) and Cmax ratio, with and without food
Module 2: Area Under Curve (AUC) | At predefined intervals throughout the treatment period (approximately 12 weeks)
  The concentration of AZD5305 in plasma will be determined. Area under the curve is the integral of the concentration-time curve. The AUC reflects the actual body exposure to drug after administration. The AUC is dependent on the rate of elimination of the drug from the body and the dose administered.
Module 2: Maximum plasma concentration of the drug (Cmax) | At predefined intervals throughout the treatment period (approximately 12 weeks)
  The concentration of AZD5305 in plasma will be determined (Cmax will be derived).
Module 2: The time taken to reach the maximum concentration (Tmax) | At predefined intervals throughout the treatment period (approximately 12 weeks)
  The concentration of AZD5305 in plasma will be determined (Tmax will be derived).
Module 3: Area Under Curve (AUC) | At predefined intervals throughout the treatment period (approximately 12 weeks)
  The concentration of AZD5305 in plasma will be determined. Area under the curve is the integral of the concentration-time curve. The AUC reflects the actual body exposure to drug after administration. The AUC is dependent on the rate of elimination of the drug from the body and the dose administered.
Module 3: Maximum plasma concentration of the drug (Cmax) | At predefined intervals throughout the treatment period (approximately 12 weeks)
  The concentration of AZD5305 in plasma will be determined (Cmax will be derived).
Module 3: The time taken to reach the maximum concentration (Tmax) | At predefined intervals throughout the treatment period (approximately 12 weeks)
  The concentration of AZD5305 in plasma will be determined (Tmax will be derived).
Module 4 : Area Under Curve | At predefined intervals throughout the treatment period (approximately 12 weeks)
  The concentration of AZD5305 in plasma will be determined. Area under the curve is the integral of the concentration-time curve. The AUC reflects the actual body exposure to drug after administration. The AUC is dependent on the rate of elimination of the drug from the body and the dose administered.
Module 4: Maximum plasma concentration of the drug (Cmax) | At predefined intervals throughout the treatment period (approximately 12 weeks)
  The concentration of AZD5305 in plasma will be determined (Cmax will be derived).
Module 4: The time taken to reach the maximum concentration (Tmax) | At predefined intervals throughout the treatment period (approximately 12 weeks)
  The concentration of AZD5305 in plasma will be determined (Tmax will be derived).
Module 4: Anti-Drug Antibody (ADA) | Samples will be collected within 1 hour before dose administration on Day 1 of Cycle 1, 2, and 4, then every 4 Cycles (each cycle is 21 days), EoT, and at safety follow-up (40 days after last dose) as per Schedule of Assessments
  To investigate the presence of ADAs for T-DXd
Module 4: To assess the preliminary anti-tumour activity of AZD5305 as monotherapy and in combination with T-DXd. | From screening to approximately 6 months
  Time from C1D1 to progression or death, as defined by RECIST v 1.1 summarised at the 6 month landmark (PFS6)
Module 5: Area Under Curve | At predefined intervals throughout the treatment period (approximately 12 weeks)
  The concentration of AZD5305 in plasma will be determined. Area under the curve is the integral of the concentration-time curve. The AUC reflects the actual body exposure to drug after administration. The AUC is dependent on the rate of elimination of the drug from the body and the dose administered.
Module 5: Maximum plasma concentration of the drug (Cmax) | At predefined intervals throughout the treatment period (approximately 12 weeks)
  The concentration of AZD5305 in plasma will be determined (Cmax will be derived).
Module 5: The time taken to reach the maximum concentration (Tmax) | At predefined intervals throughout the treatment period (approximately 12 weeks)
  The concentration of AZD5305 in plasma will be determined (Tmax will be derived).
Module 5: Anti-Drug Antibody (ADA) | Whole blood samples for determination of ADA for Dato-DXd in plasma will be collected in patients receiving Dato-DXd per the schedule specified in the SoA : Day 1 of Cycle 1, 2, 4, and 8 (each cycle is 21 days) , EoT, and then 28 day follow up visit.
  Presence of ADAs for Dato-DXd
Module 5: Premilinary anti tumour activity AZD5305 in combination with Dato-DXd | From screening to confirmed progresive disease ( approximately 12 weeks)
  objective response rate and radiographic progression-free survival using RECIST v1.1.
  Proportion of patients achieving a ≥ 50% decrease in PSA from baseline to the post-baseline PSA result, confirmed by a second consecutive PSA assessment at least 3 weeks later (PSA50 response).
Module 6: To characterise the PK of AZD5305 and camizestrant following a single dose and at steady state after multiple dosing, when given in combination. | At predefined interval throughout the treatment (approximately 12 weeks)
  Plasma concentrations and PK parameters of AZD5305 and camizestrant after single dose and multiple dose administration, including, but not limited to:
  AUC, Cmax, Tmax, as data allow
Module 6: To evaluate the effect of camizestrant on the PK of AZD5305. | At predefined intervals throughout the treatment period (approximately 12 weeks)
  PK parameters, including but not limited to AUC and/or AUC(0-t), Cmax, Tmax, AUC(0-t) and Cmax ratio, with and without camizestrant.
Module 6: To evaluate the effect of AZD5305 on the PK of Camizestrant. | At predefined intervals throughout the treatment period (approximately 12 weeks)
  PK parameters, including but not limited to AUC and/or AUC(0-t), Cmax, Tmax, AUC(0-t) and Cmax ratio, with and without AZD5305.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Yap, Principal Investigator — M.D. Anderson Cancer Center
Locations (54):
- United States (4):
  - Research Site, Boston, Massachusetts
  - Research Site, New York, New York
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Houston, Texas
- Australia (2):
  - Research Site, Heidelberg
  - Research Site, Melbourne
- Canada (3):
  - Research Site, Vancouver, British Columbia
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- China (13):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Harbin
  - Research Site, Jining
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Taiyuan
  - Research Site, Wuhan
  - Research Site, Xi'an
- Czechia (2):
  - Research Site, Brno
  - Research Site, Prague
- Research Site, Budapest, Hungary
- Italy (5):
  - Research Site, Milan
  - Research Site, Modena
  - Research Site, Napoli
  - Research Site, Padua
  - Research Site, Roma
- Japan (2):
  - Research Site, Chūōku
  - Research Site, Kōtoku
- Poland (7):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Grzepnica
  - Research Site, Lodz
  - Research Site, Torun
  - Research Site, Warsaw
- Research Site, Moscow, Russia
- Research Site, Seoul, South Korea
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pozuelo de Alarcón
  - Research Site, Seville
- Ukraine (4):
  - Research Site, Chernivtsі
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Uzhhorod
- United Kingdom (4):
  - Research Site, Cambridge
  - Research Site, Manchester
  - Research Site, Oxford
  - Research Site, Sutton

REFERENCES:
- [Derived] Illuzzi G, Staniszewska AD, Gill SJ, Pike A, McWilliams L, Critchlow SE, Cronin A, Fawell S, Hawthorne G, Jamal K, Johannes J, Leonard E, Macdonald R, Maglennon G, Nikkila J, O'Connor MJ, Smith A, Southgate H, Wilson J, Yates J, Cosulich S, Leo E. Preclinical Characterization of AZD5305, A Next-Generation, Highly Selective PARP1 Inhibitor and Trapper. Clin Cancer Res. 2022 Nov 1;28(21):4724-4736. doi: 10.1158/1078-0432.CCR-22-0301. PMID 35929986
- See also: Breast Cancer Study Locator details (for US) — https://www.breastcancerstudylocator.com/trial/listing/260668